CLINICAL TRIAL: NCT01157793
Title: A Multicentre, Randomised, Open-label, Controlled Study to Evaluate the Effects of Saizen® on Cardiac Function in GHD Subjects During the Transition Phase From Childhood to Adulthood
Brief Title: A Multicentre, Randomised, Open-label, Controlled Study to Evaluate the Effects of Saizen® on Cardiac Function in Growth Hormone Deficient(GHD) Subjects During the Transition Phase From Childhood to Adulthood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sonia Shin, Head of Medical Department, Merck Serono Korea, an affiliate of MerckKGaA, Darmstadt, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP24632
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2010-07

CONDITIONS: Dwarfism; Growth Hormone Deficiency
Keywords: Dwarfism; Growth hormone deficiency; Growth hormone
MeSH Terms: conditions — Dwarfism; Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: r-hGH
- Group 2 (Experimental)
  Interventions: Drug: r-hGH

INTERVENTIONS:
Drug: r-hGH — r-hGH at a dose of 0.15-1.00 mg/day administered for 48 weeks by s.c. route
  Other Names: Saizen®
  Arms: Group 1
Drug: r-hGH — Initially no treatment for the first 24 weeks followed by administration of r-hGH at a dose of 0.15 1.00 mg/day for the next 24 weeks, by s.c. route
  Other Names: Saizen®
  Arms: Group 2

SUMMARY:
This was a 48-week, open-label, prospective, multicentric, randomised, comparative with parallel control, Phase 4 study to evaluate the effects of Saizen on cardiac function in GHD subjects during the transition phase from childhood to adulthood.

The study was designed to evaluate whether recombinant-human growth hormone (r-hGH) treatment also benefits young subjects with GHD. Some trials have already been published on this subject, but they were mainly focused on the bone density.

DETAILED DESCRIPTION:
Growth hormone is a 191 amino acid polypeptide hormone (MW 22,000) normally synthesised and secreted by the somatotrophic cells of the anterior lobe of the pituitary gland. In normal development, growth hormone and somatomedins are responsible for many of the manifestations of normal growth and GHD is manifested by a marked short stature. Growth hormone deficiency has been treated by human growth hormone for many years. Serono's r-hGH (Saizen) is produced from genetically engineered mammalian cells.

The findings from previous clinical studies on GH treatment in GH-deficient adults, collectively indicate that the majority of adults with long-standing GH deficiency, whether dating from childhood or acquired in adult life, are compromised both physically and psychologically and can derive clinical benefit from GH replacement. Based on observations in the clinical trials to date , a GH dose of 0.01 mg/kg/day (50% of the dose used in children), is likely to be satisfactory for many subjects. Moreover, it should be possible to minimise early side effects, particularly fluid retention, by initiating treatment with half of this dose and increasing to the final dose after 4 weeks if well tolerated.

In this study, it was proposed to enroll a group of childhood onset GHD subjects who were not treated with r-hGH. Half of the study population started treatment for six months whilst the other half remained on no r-hGH treatment. After six months the group already on r-hGH therapy continued treatment for a further six months and the second group presently on no r-hGH treatment started r hGH treatment for the remaining six months of the study.

OBJECTIVES

Primary objective:

* To compare the effects of Saizen on cardiac function (as assessed by percentage ejection fraction) in subjects where 50% of the study population started r-hGH treatment for 24 weeks and then remained on r-hGH treatment for a further 24 weeks and subjects who continued on no r-hGH for 24 weeks before starting r-hGH for 24 weeks during the transition phase from childhood to adulthood.

Secondary objectives:

- To assess the safety and tolerability of r-hGH in subjects who were transitioning from childhood to adulthood, and to assess the change in body composition and lean body mass. Subsidiary analyses of the other echocardiography parameters was also performed.

After entry into the trial, the subjects were randomised to one of two groups for a 48-week period:

* Group 1: Saizen (r-hGH), 0.15-1.00 mg/day for 48 weeks, subcutaneous (s.c.)
* Group 2: No treatment for the first 24 weeks followed by Saizen (r-hGH)0.15-1.00 mg/day for the next 24 weeks, s.c.

Subjects' visits to the study site was scheduled as follows:

* Group 1 - Baseline (study day 1), weeks 4, 12, 24, 36 & 48.
* Group 2 - Baseline (study day 1), weeks 12, 24, 28, 36 & 48. The study drug was administered subcutaneously once daily in the evenings during the active treatment period. The dose was to be adjusted stepwise, controlled by Insulin-Growth Factor-I (IGF-I) values. The recommended final r-hGH dose was not to exceed 1.00mg/day

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of childhood onset GH deficiency and previously treated with GH
* Subjects who had attained final height
* Male or female subjects, aged between 14 and 25 years of age inclusively at baseline
* Subjects with GH deficiency of <5μg/L (acquired or idiopathic), established by any 1 type of GH secretion test within 3 years prior to Study Day 1
* If hypopituitary, subject must have been on adequate replacement therapy (if required) of glucocorticosteroids, thyroid & sex hormones (hormones levels on replacement being in normal/mildly elevated range) for at least 6 months prior to study entry
* Subjects who were willing and able to comply with the protocol for the duration of the study.
* Subjects who had given written informed consent before any study-related procedure not part of the subject's normal medical care, with the understanding that the subject might withdraw consent at any time without prejudice to future medical care
* Female subjects must be neither pregnant nor breast-feeding, and use a hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Confirmation that a female subject was not pregnant was established by a negative urinary human chorionic gonadotropin (hCG) pregnancy test at baseline.

Exclusion Criteria:

* Subject who had a known allergy or hypersensitivity to growth hormone or diluent
* Subject who had been treated with r-hGH in previous six months
* Subject with chronic severe kidney disease
* Subject with chronic severe liver disease
* Subject with acute or severe illness during the previous 6 months
* Subject with significant concomitant illness which would interfere with his/her participation or assessment in this study
* Subject with active malignancy (except non-melanomatous skin malignancies)
* Subjects with unstable hypertension (supine systolic blood pressure persistently above 160 mmHg or diastolic blood pressure persistently above 100 mmHg)
* Subjects with benign cranial hypertension
* Subjects with a history of carpal tunnel syndrome, unless surgically released
* Subjects with known positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) and/or Hepatitis C virus (HCV) serology based on past medical history
* Subjects with known active drug addiction, including alcoholism, or use of drugs for nontherapeutic purposes
* Subject who had previously participated in this study
* Subject taking an investigational drug or enrolled in another clinical study

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2003-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change in percentage ejection fraction in subjects during the transition phase from childhood to adulthood | Baseline to study week 48

SECONDARY OUTCOMES:
Subsidiary analysis of the other echocardiography parameters and lean body mass | Baseline to study week 48
Evaluation of laboratory parameters and monitoring of adverse events | Baseline to study week 48

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Wee, MD, Study Director — Merck Serono International SA